CLINICAL TRIAL: NCT07328984
Title: How Long Should we Give Steroids for Patients With Severe PCP (HOW LONG)
Brief Title: How Long Should we Give Steroids for Patients With Severe PCP
Acronym: HOW LONG
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Emily McDonald, Associate professor of medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2026-12265; 527077 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Pneumocystis Pneumonia; Pneumocystis; Pneumocystis Jirovecii Infection; Pneumocystis Jiroveci Pneumonia; Pneumocystis Carinii; Infection, Resulting From HIV Disease; Pneumocystosis Associated With AIDS; Pneumocystosis; Pneumonia (Etiology)
Keywords: PCP; Systemic Corticosteroids; De-escalation of Therapy; Randomized Control Trial; Immunocompromised host; HIV; Non-HIV; Pneumocystis jirovecii pneumonia
MeSH Terms: conditions — Pneumonia, Pneumocystis; Pneumocystis Infections; Infections; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shortened-Duration Corticosteroids (Experimental): Discontinue adjunctive systemic corticosteroids at day 10 of therapy or at hospital discharge (whichever occurs first), after documented clinical recovery (room air for ≥6 hours).
  Interventions: Drug: Systemic corticosteroids
- Standard duration of Corticosteroids (Active Comparator): Continue adjunctive systemic corticosteroids to a total of 21 days (standard of care).
  Interventions: Drug: Systemic corticosteroids

INTERVENTIONS:
Drug: Systemic corticosteroids — Adjunctive systemiccorticosteroid therapy administered as part of standard treatment for pneumocystis Pneumonia, with duration varying by study arm.

SUMMARY:
The HOW LONG trial is an international, multicenter, Phase IV randomized clinical trial evaluating the optimal duration of adjunctive systemic corticosteroids in immunocompromised adults with severe Pneumocystis jirovecii pneumonia (PCP) who demonstrate early clinical recovery. Participants who no longer require supplemental oxygen by day 10 of corticosteroid therapy are randomized to discontinue corticosteroids at day 10 (or hospital discharge, if earlier) versus continue corticosteroids for a total of 21 days. The trial assesses whether earlier discontinuation reduces steroid-related complications while maintaining clinical outcomes.

DETAILED DESCRIPTION:
Adjunctive systemic corticosteroids are routinely used in severe PCP to reduce pulmonary inflammation and improve survival, but the recommended 21-day duration is based on limited historical evidence. Prolonged corticosteroid exposure may increase risks including secondary infections, hyperglycemia, gastrointestinal bleeding, and other adverse effects. The HOW LONG trial tests whether stopping corticosteroids earlier, after clinical recovery, improves net clinical outcomes.

Eligible adults with proven or probable severe PCP who have recovered to room air (no need for supplemental oxygen) for at least 6 hours by day 10 of corticosteroid therapy are enrolled and randomized centrally 1:1 in the MUHC Research Electronic Data Capture (REDCap) system to (1) discontinuation of corticosteroids at day 10 or hospital discharge or (2) continuation of corticosteroids to a total of 21 days. All participants receive standard antimicrobial therapy for PCP per treating clinicians. Follow-up occurs to day 180.

The primary endpoint is a hierarchical composite outcome assessed at day 60, incorporating mortality, relapse of PCP-related hypoxemia, secondary infections, severe metabolic or gastrointestinal complications, and length of hospital stay. Secondary endpoints include individual components of the composite outcome, and tertiary endpoints include quality of life and longer-term outcomes through day 180.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Proven or probable Pneumocystis jirovecii pneumonia
* Severe PCP requiring supplemental oxygen (e.g., ≥4 L/min or ≥35% FiO₂ to maintain SpO₂ ≥94%)
* Planned or receiving adjunctive systemic corticosteroid therapy for severe PCP
* Clinical recovery by day 10 of steroid therapy: breathing room air for ≥6 hours
* Able to provide informed consent (or per local requirements)

Exclusion Criteria:

* Persistent hypoxemia or ongoing oxygen requirement at day 10
* Clinical deterioration prior to randomization
* Treating clinician determines steroids must be continued or stopped immediately for medical reasons
* Anticipated death within 48 hours
* Inability or unwillingness to complete follow-up through day 180

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite clinical outcome | Day 60
  The primary outcome at day 60 will be the hierarchical composite of:
  1. death,
  2. relapse of PCP-related hypoxemia (e.g., not due to another obviously identified cause like pulmonary embolism, aspiration event, etc.) requiring more than 12 hours of use of ≥2L of oxygen in accordance with guidelines
  3. The development of secondary infections requiring systemic antibiotic therapy
  4. The development of severe diabetic complications (ketoacidosis, hyperosmolar coma, new initiation of insulin which is continued at discharge)
  5. The development of severe GI bleeding (e.g., necessitating unplanned transfusion and/or endoscopy) and;
  6. inpatient length of stay (censored at day 60; deaths assigned 60 days).

SECONDARY OUTCOMES:
Death | Day 60
  Mortality at day 60
relapse of PCP-related hypoxemia | Day 60
  (Relapse of PCP-related hypoxemia that is not due to another obviously identified cause like pulmonary embolism, aspiration event, etc.) requiring more than 12 hours of use of ≥2L of oxygen in accordance with guidelines
Secondary infections requiring systemic antibiotic therapy | Day 60
  The development of secondary infections requiring systemic antibiotic therapy
The development of severe diabetic complications | Day 60
  Severe complications of diabetes include: ketoacidosis, hyperosmolar coma, new initiation of insulin which is continued at discharge
The development of severe GI bleeding ( | Day 60
  Gastrointestinal bleeding necessitating unplanned transfusion and/or endoscopy
inpatient length of stay (censored at day 60; deaths assigned 60 days). | Day 60
  inpatient length of stay censored at day 60; deaths assigned 60 days.

OTHER OUTCOMES:
Quality of life (EQ-5D-5L) | Day 30
  Higher score indicates better quality of life
Quality of life (EQ-5D-5L) | Day 180
  Higher score indicates better quality of life
All-cause mortality | Day 180
  all cause mortality
PCP recurrence | Day 180
  recurrence of PCP infection following the initial infection

CONTACTS AND LOCATIONS:
Locations (1):
- McGill university Health Centre (Royal victoria Hospital and Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available upon reasonable request to the principal investigator by email (emily.mcdonald@mcgill.ca) subject to discussion surrounding the necessity of an interinstitutional data sharing agreement, commencing one year following the publication of the main trial results, for a period of 2 years.
Time Frame: 1 year following main publication for a period of 2 years
Access Criteria: investigators wishing to pursue secondary questions related to the data can contact emily.mcdonald@mcgill.ca for access to the data via a data sharing agreement.

REFERENCES:
- [Background] Senecal J, Smyth E, Del Corpo O, Hsu JM, Amar-Zifkin A, Bergeron A, Cheng MP, Butler-Laporte G, McDonald EG, Lee TC. Non-invasive diagnosis of Pneumocystis jirovecii pneumonia: a systematic review and meta-analysis. Clin Microbiol Infect. 2022 Jan;28(1):23-30. doi: 10.1016/j.cmi.2021.08.017. Epub 2021 Aug 28. PMID 34464734
- [Background] McDonald EG, Butler-Laporte G, Del Corpo O, Hsu JM, Lawandi A, Senecal J, Sohani ZN, Cheng MP, Lee TC. On the Treatment of Pneumocystis jirovecii Pneumonia: Current Practice Based on Outdated Evidence. Open Forum Infect Dis. 2021 Oct 29;8(12):ofab545. doi: 10.1093/ofid/ofab545. eCollection 2021 Dec. PMID 34988242